CLINICAL TRIAL: NCT04242797
Title: Central Mechanisms of Calmare: an fMRI Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Collaborators: Sorenson Legacy Foundation (Unknown); Brigham Young University MRI Research Facility (Unknown)
Responsible Party: Principal Investigator, David D Busath, Professor, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F15130
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Neuropathy
Keywords: Idiopathic; diabetic; chemotherapy-induced
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Equal numbers of participants are randomly assigned to either the Calmare or traditional TENS group. Using skin electrodes positioned by the therapist proximal to the limb pain, each participant is given the assigned stimulation mode for 30-minute therapy sessions. One therapy is used in the pilot study and ten therapies on consecutive weekdays in the extended study.
Who Masked: Participant, Care Provider
Masking Description: The investigator uses Bluetooth to control the output of a switching box for each patient from outside the treatment room. The box controls whether the inputs from the Calamare device or two traditional dual-channel TENS devices are connected to the output. The stimulus amplitude knobs for the TENS units are ganged to those of the Calmare using O-rings. When the therapist increases the stimulus amplitude on Calmare, that of the corresponding TENS unit is increased to about the same extent simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Calmare (Active Comparator): Single- or ten-dose treatments on consecutive weekdays, 30 minutes each.
  Interventions: Device: Calmare
- Traditional TENS (Active Comparator): Single- or ten-dose treatments on consecutive weekdays, 30 minutes each.
  Interventions: Device: TENS

INTERVENTIONS:
Device: Calmare — Skin is stimulated with an electrical voltage via electrode pads, variably distorted sine wave at ~47 Hz.
  Arms: Calmare
Device: TENS — Skin is stimulated with an electrical voltage via electrode pads, 300 micro-second rectangle pulse at 47 Hz.
  Other Names: Traditional TENS
  Arms: Traditional TENS

SUMMARY:
Pilot one-treatment and extended 10-treatment studies are carried out on participants with peripheral neuropathy comparing traditional TENS and Calmare stimulation protocols using a double-blind apparatus. Resting fMRI scans are obtained before and after the treatment, as well as after most of the pain has returned.

DETAILED DESCRIPTION:
Pain can be either useful or harmful. Acute pain conveys information to the brain about real or potential damage that can productively lead to avoidance or treatment of the damage. However, chronic pain, which extends beyond these useful purposes, becomes a potentially debilitating inconvenience. Estimations based on surveys report that as many as 33% of Americans suffer from chronic pain, with a significant portion being unable to successfully manage it.

The current means to treating chronic pain include: surgery, drug therapy, physical therapy, psychological intervention, and others. Unfortunately, despite these options, many people continue to suffer from a chronic pain condition. Neuropathic pain, or pain caused by nervous system damage, is particularly hard to treat. Drug therapy and surgery have relatively low success rates and undesirable side effects. Thus, there is a need for additional research and new treatment methods for neuropathic pain patients.

The Calmare device was designed as one such means to treat chronic neuropathic pain. It works through electrostimulation of the skin near the pain site, and, according to recent studies, has significantly reduced chronic neuropathic pain in most subjects (Majithia et al., 2016).

Previous studies of Calmare effectiveness have defined the success of treatment as the reduction of reported pain levels by the patient. Though useful, these studies fail to provide an objective measurement of pain reduction and fail to discover the mechanisms by which it occurs. In addition, previous studies have been unable to perform a true double-blind experiment in which the placebo effect was entirely accounted for. The pilot study takes a step toward filling this gap by performing a double blind, randomized single-treatment trial comparing Calmare efficacy to traditional transcutaneous electrical nerve stimulation (TENS) efficacy. The ten-treatment study examines the durability of the pain relief for 12 weeks after the treatment period.

The goal of these studies is two-fold: first, to use fMRI before and after a full therapeutic Calmare treatment course to determine the extent to which Calmare affects the connectivity of the pain centers of the brain, and second, to determine whether traditional TENS or Calmare is more effective in reducing neuropathic chronic pain. The Calmare treatment is administered in a double-blind fashion with neither the technician, nor the subject knowing whether the TENS or the Calmare is being administered. The investigator's hypothesis is that Calmare therapy decreases subject pain through a central mechanism that will be manifest in decreased functional connectivity of the brain's pain centers. The degree to which this happens is determined by comparing the decrease in pain intensity, as reported by the patient, with the difference in fMRI BOLD temporal correlations between pain centers.

ELIGIBILITY:
Inclusion Criteria:

* They must have suffered from a diagnosed peripheral neuropathy (diabetic, chemotherapy induced, or other) for a minimum of 6 months.
* At the time of the study they must experience pain greater than or equal to 5 on a visual analog pain scale from 0-10, with 0 being "no pain" and 10 being "the worst imaginable pain."

Exclusion Criteria:

* pregnancy
* a history of epilepsy or brain damage
* presence of a serious psychiatric disorder (e.g. schizophrenia, manic-depressive psychosis, primary major depression)
* multiple sources of chronic pain (e.g. a chronic pain condition other than a peripheral neuropathy or more than one site of neuropathies)
* a skin condition that would prevent application of skin electrodes
* latex allergy
* severe arrhythmia or any form of equivalent heart disease
* history of myocardial infarction or ischemic heart disease within the past 6 months
* celiac plexus block or other neurolytic pain control treatment within the past 4 weeks
* state of active withdrawal from drugs and/or alcohol
* ineligible for fMRI due to metal implants, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Visual Analaog Scale (VAS) Pain Score Changes | The intra-subject change in VAS score from pre-Rx baseline a) after the 30-minute treatment and b) again the next day (pilot), or a) after each of the ten 30-minute treatments and b) 6- and 12-weeks from end of treatment (extended)
  Change from baseline in VAS score, which is marked on a line labeled 0 on the left (no pain) and 10 on the right (the most exquisite pain imaginable).
Washington Neuropathic Pain Scale (WNPS) Pain Score Changes | The intra-subject change in ten WNPS pain scores from baseline after the 30-minute Rx and again the next day (pilot) or after each of the ten 30-minute Rxs and 6- and 12-weeks from end of Rx period (extended)
  Change from baseline in each of ten WNPS scores, which are marked boxes have integral values of 0 on the left (no pain) and 10 on the right (the most exquisite pain imaginable).
Changes in resting fMRI Correlations | Intra-subject changes in fMRI signals from baseline (taken immediately before first Rx) obtained 30 minutes after first Rx (pilot) or 10th Rx (extended) and again 24 hours later (pilot) or 6-weeks later (extended).
  Change in temporal correlations of resting fMRI signals from 93 cerebral regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: David D Busath, M.D., Principal Investigator — Brigham Young University
Locations (1):
- BYU MRI Research Facility, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majithia N, Smith TJ, Coyne PJ, Abdi S, Pachman DR, Lachance D, Shelerud R, Cheville A, Basford JR, Farley D, O'Neill C, Ruddy KJ, Sparadeo F, Beutler A, Loprinzi CL. Scrambler Therapy for the management of chronic pain. Support Care Cancer. 2016 Jun;24(6):2807-14. doi: 10.1007/s00520-016-3177-3. Epub 2016 Apr 4. PMID 27041741

DOCUMENTS (1):
  • Informed Consent Form (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04242797/ICF_000.pdf